CLINICAL TRIAL: NCT02105532
Title: A Multi-centre, Feasibility, Cluster Randomised Controlled Trial Comparing Restrictive Versus Liberal Blood Transfusion Strategies in Adult Patients Admitted With Acute Upper Gastrointestinal Bleeding
Brief Title: Transfusion in Gastrointestinal Bleeding
Acronym: TRIGGER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr Vipul Jairath (Other Government)
Collaborators: NHS Blood and Transplant (Other Government)
Responsible Party: Sponsor-Investigator, Dr Vipul Jairath, Research Fellow in Gastroneterology, NHS Blood and Transplant
Organization: NHS Blood and Transplant (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-09-CSU; ID 12078 (Other: NIHR)
Record Dates: First submitted 2012-07-24; First posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Gastrointestinal Hemorrhage
Keywords: Transfusion in gastrointestinal bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Restrictive Transfusion Policy (Active Comparator): Participants allocated to this group will be eligible for transfusion once their Hb level is ≤ 8 g/dL after presentation to hospital. The objective for the attending clinician is to maintain the Hb level between 8.1-10 g/dL for the duration of hospital stay.
  Interventions: Other: Restrictive transfusion policy
- Liberal Transfusion Policy (Active Comparator): Participants allocated to this group will be eligible for transfusion once their Hb level is ≤ 10 g/dL after presentation to hospital. The objective for the attending clinician is to maintain the Hb level between 10.1-12 g/dL for the duration of hospital stay.
  Interventions: Other: Liberal Transfusion Policy

INTERVENTIONS:
Other: Restrictive transfusion policy — Participants allocated to this group will be eligible for transfusion once their Hb level is ≤ 8 g/dL after presentation to hospital. The objective for the attending clinician is to maintain the Hb level between 8.1-10 g/dL for the duration of hospital stay.
  Arms: Restrictive Transfusion Policy
Other: Liberal Transfusion Policy — Participants allocated to this group will be eligible for transfusion once their Hb level is ≤ 10 g/dL after presentation to hospital. The objective for the attending clinician is to maintain the Hb level between 10.1-12 g/dL for the duration of hospital stay.
  Arms: Liberal Transfusion Policy

SUMMARY:
Aim: To evaluate the feasibility and safety of a restrictive versus liberal red blood cell (RBC) transfusion policy in adult patients admitted with Acute Upper Gastrointestinal Bleeding (AUGIB) in order to inform the design of a definitive phase III randomised controlled trial.

DETAILED DESCRIPTION:
Trial overview: TRIGGER is a pragmatic trial aiming to recruit adult patients admitted with all cause AUGIB (non-variceal and variceal). The study will take place in six United Kingdon hospitals and they will be randomly allocated to a transfusion policy at the cluster level; three sites will be allocated to a restrictive transfusion policy and three to a liberal transfusion policy. Given the challenges that will be involved in early recruitment and cross-speciality care, a feasibility study is essential to determine whether a sufficient proportion of eligible patients can be recruited into the trial and that clinicians can adhere to the allocated transfusion policy. Recruitment will operate for 6 months in total. The investigators will compare recruitment rate, protocol adherence, clinical characteristics of patients recruited, exposure to RBC transfusions and the difference in Hb concentrations between the restrictive and liberal transfusion policies. The investigators will collect important clinical outcomes which the investigators anticipate being central to the phase III trial, including 28-day mortality, further bleeding rates and serious adverse events between the restrictive and liberal transfusion policies. The investigators will also collect data to enable us to plan a health economic evaluation and quality of life assessment for the phase III trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or over years presenting with AUGIB, defined by haematemesis or melaena.

Exclusion Criteria:

* Patients with whom the responsible clinician considers there is a need for immediate RBC transfusion prior to obtaining or regardless of the initial Hb result due to severity of bleeding.
* Existing hospital in-patients who develop AUGIB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 936 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Adherence to the study protocol | up to 28 days
  Protocol adherence will be measured over time, to determine if adherence rates improve. Adherence rates will also be compared between transfusion arms.

SECONDARY OUTCOMES:
Further Bleeding | up to 28 days
  Further bleeding up to Day 28: Further bleeding is a composite outcome that includes persistent bleeding (defined as any bleeding present at the end of the index endoscopy, regardless of whether endoscopic therapy was attempted or not), and recurrent bleeding. Recurrent bleeding is only assessed in patients without persistent bleeding, and must be confirmed by the presence of high-risk stigmata of bleeding either endoscopically, radiologically, or surgically. Recurrent bleeding should initially be suspected in the event of any combination of the following: fresh haematemesis, continuous melaena, or aspiration of fresh blood from a naso-gastric tube, with a pulse rate of >100 bpm, a fall in systolic blood pressure of >30mm Hg or a drop in Hb of >2g/dL in the preceding 24 hours. Persistent bleeding and recurrent bleeding will also be assessed separately.

OTHER OUTCOMES:
Red Blood Cell exposure in patients | up to 28 days
  The difference in number of red blood cell units administered will be compared between the intervention groups up to discharge/death/Day 28 (whichever comes first).
Selection bias | 6 months
  Clinical characteristics of patients in the two transfusion policies
Difference in Hb concentration Between Restrictive and Liberal Groups | up to 28 days
  The mean Hb values for patients will be compared between the treatment arms up to discharge/death/Day 28 (whichever comes first).
Death | up to 28 days
  All-cause mortality up to Day 28.
Need for therapeutic intervention at the index endoscopy | up to 28 days
  This includes any therapeutic modality performed for AUGIB at the index endoscopy.
Need for surgery or radiological intervention to control bleeding | up to 28 days
Proportion of patients experiencing the composite endpoint of thromboembolic and ischaemic events up to Day 28 | up to 28 days
  Includes myocardial infarction, stroke, pulmonary embolus, Deep Vein Thrombosis, acute kidney injury. Each component will also be assessed individually. See section 8.1.3 for a definition of ischaemic and thromboembolic events.
Acute Transfusion reactions up to death/ discharge | up to 28 days
  Defined as a reaction occurring at any time up to 24 hours following a transfusion of a blood component.
Infections | up to 28 days
  Any infection necessitating a prescription for the use of antibiotic treatment for a minimum of 5 days, provided the prescription is received before or on Day 28.
Length of hospital stay | up to 28 days
Health related quality of life at Day 28 | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Professor Michael F Murphy, Study Chair — NHS Blood and Transplant; Vipul Jairath, Study Director — NHSBT and Translational Gastroenterology Unit, Oxford, UK.
Locations (1):
- NHSBT Clinical Studies Unit, Oxford, United Kingdom

REFERENCES:
- [Derived] Kahan BC, Jairath V. Outcome pre-specification requires sufficient detail to guard against outcome switching in clinical trials: a case study. Trials. 2018 May 2;19(1):265. doi: 10.1186/s13063-018-2654-z. PMID 29720248
- [Derived] Jairath V, Kahan BC, Gray A, Dore CJ, Mora A, James MW, Stanley AJ, Everett SM, Bailey AA, Dallal H, Greenaway J, Le Jeune I, Darwent M, Church N, Reckless I, Hodge R, Dyer C, Meredith S, Llewelyn C, Palmer KR, Logan RF, Travis SP, Walsh TS, Murphy MF. Restrictive versus liberal blood transfusion for acute upper gastrointestinal bleeding (TRIGGER): a pragmatic, open-label, cluster randomised feasibility trial. Lancet. 2015 Jul 11;386(9989):137-44. doi: 10.1016/S0140-6736(14)61999-1. Epub 2015 May 5. PMID 25956718
- [Derived] Campbell HE, Stokes EA, Bargo D, Logan RF, Mora A, Hodge R, Gray A, James MW, Stanley AJ, Everett SM, Bailey AA, Dallal H, Greenaway J, Dyer C, Llewelyn C, Walsh TS, Travis SP, Murphy MF, Jairath V; TRIGGER investigators. Costs and quality of life associated with acute upper gastrointestinal bleeding in the UK: cohort analysis of patients in a cluster randomised trial. BMJ Open. 2015 Apr 29;5(4):e007230. doi: 10.1136/bmjopen-2014-007230. PMID 25926146